CLINICAL TRIAL: NCT01164345
Title: Plerixafor (Plerixafor AMD 3100) + Recombinant Human G-CSF (rhG-CSF) for Autologous Peripheral Blood Stem Cell Transplantation (AutoSCT) in Hard to Mobilise Patients: a Phase IIB Study
Brief Title: Mozobil for Autologous Stem Cell Mobilization
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-09-7481-AN-CTIL
Record Dates: First submitted 2010-07-12; First posted 2010-07-16 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Non-Hodgkin's Lymphoma; Hodgkin's Lymphoma; Stem Cell Mobilization; Autologous Stem Cell Transplantation
Keywords: non-Hodgkin's lymphoma; Hodgkin's lymphoma; stem cell mobilization; autologous stem cell transplantation
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease | interventions — plerixafor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MOZOBIL (Experimental): treatment with mozobil for autologous stem cell collection
  Interventions: Drug: Plerixafor

INTERVENTIONS:
Drug: Plerixafor — Plerixafor (mozobil) 240 mcg/kg SC will be administered in the evening, 10 hours prior to initiation of apheresis.G-CSF will be administered in the morning at 10 mcg/kg SC for 4 days prior to apheresis.
  Other Names: Mozobil and Neupogen

SUMMARY:
The aim of this study is to evaluate Plerixafor (MOZOBIL) plus recombinant human G-CSF (G-CSF) efficiency in mobilizing sufficient number of stem cells from Lymphoma (NHL and HL) patients for autologous transplantation.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible and planned for an autologous haematopoietic stem cell transplantation.

1.1 Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.

1.2 WBC count ≥2.5x109/L.

1.3 Absolute neutrophil count ≥1.5x109/L.

1.4 Platelet count ≥100x109/L

1.5 Adequate cardiac, renal, hepatic and pulmonary function sufficient to undergo apheresis and transplantation.

1.6 Previously, heavily pretreated lymphoma patients or patients suspected to have a poor bone marrow stem cell reserve for at least one of the following:

* >2 lines of chemotherapy.
* Previous radiotherapy involving bone marrow
* Prior therapy with specific stem cell toxic chemotherapeutic agents
* Platelets count pre-mobilisation, ≤150.103 x mm3
* Level of circulating CD34+ ≤ 20 cells/mcL prior to apheresis on the collection day
* Patients > 60 years of age

Exclusion Criteria:

2.1 Lymphoma patients that did not fulfil the inclusion criteria.

2.2 History of any acute or chronic leukemia (including myelodysplastic syndrome.

2.3 Prior allogeneic or autologous transplantation.

2.4 Inability to tolerate stem cell harvest.

2.5 Peripheral venous access not possible.

2.6 Pregnant or nursing women.

2.7 Positive serology for hepatitis B or C.

2.8 Acute infection (febrile, i.e. temperature > 38C) within 24 hours prior to dosing or antibiotic therapy within 7 days prior to the first dose of GCSF.

2.9 HIV positive.

2.10 Left ventricular ejection fraction < 50%.

2.11 DLCO < 50%.

2.12 Splenectomised or splenic irradiation.

2.13 Psychiatric, addictive, or any disorder/disease which compromises ability to give informed consent for participation in this study.

2.14 Treatment with other investigational drugs within 4 weeks of enrolling in this protocol or currently enrolled in another investigational protocol during the mobilisation phase.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Mobilisation success rate | 4 weeks
  Mobilisation success rate is defined as the mobilisation of a PBSC graft containing >2x106 CD34+ cells/kg in ≤ 4 apheresis sessions. We will evaluate the time from chemotherapy to stem cell collection,number of collections required to reach >2x106 CD34+ cells/kg, number of CD34+ cells collected and percentage of patients reaching >5x10 CD34+ cells/kg in ≤ 4 apheresis sessions.

SECONDARY OUTCOMES:
engraftment after transplantation | 100 days
  speed of engraftment is determined by the time until recovery of blood counts after transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Nagler, MD, Principal Investigator — Chaim Sheba Medical Center
Locations (1):
- Chaim Sheba Medical Center, Tel Litwinsky, Israel